CLINICAL TRIAL: NCT07372235
Title: Comparison at Overweight Between Those Who Receive Feedback Concerning Their Metabolic Profile or Not During an Intervention With Modified Starch- and Sucrosereduced Diet (SSRD)
Brief Title: SSRD and Overweight
Acronym: SSRD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Region Skåne FoUU (Unknown)
Responsible Party: Principal Investigator, Bodil Ohlsson, Professor, Region Skane
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-07349-01
Record Dates: First submitted 2026-01-08; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Overweight (BMI > 25)
Keywords: overweight; SSRD; metabolomics; feedback on dietary efficiency
MeSH Terms: conditions — Overweight | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary intervention without feedback (Active Comparator): All participants in this arm will be recommended SSRD, but they do not receive any information about changes in their metabolic profiles after the 6-week control
  Interventions: Other: Dietary intervention with SSRD without any feedback on metabolic profile
- Dietary intervention with feedback (Active Comparator): All participants in this arm will be recommended SSRD, and they receive information about changes in their metabolic profiles after the 6-week control
  Interventions: Other: Dietary intervention with SSRD in combination with feedback information about the metabolic profile

INTERVENTIONS:
Other: Dietary intervention with SSRD in combination with feedback information about the metabolic profile — All participants will recieve a dietary intervention. They will be informed at the 6-week control about the changes in metabolic profile since study start.
  Arms: Dietary intervention with feedback
Other: Dietary intervention with SSRD without any feedback on metabolic profile — All particpants will receive informaiton about the SSRD diet. However, the participants will not be informed about the metabolic profile at the 6-week control
  Arms: Dietary intervention without feedback

SUMMARY:
The investigators have previously found that a starch- and sucrosereduced diet (SSRD) has led decreased gastrointestinal symptoms in patients with irritabel bowel syndrome (IBS). At the same time, investigators found that the weight was reduced and the nutrient intake was improved with a more favorable metabolic profile. However, it is a challenge to change lifestyle, and most persons fail to keep on with an improved diet for a long time. Investigators therefore now want to conduct a clinical trial with SSRD in overweight/obesity for 3 months. Persons with a BMI >25 kg/m2 will be included. To examine whether a feedback about improved metabolic profile enhances the compliance, participants will be randomized to be informed or not about the metabolic profile after the 6-week visit. Investigator´s hypothesis is that information about the improvement in the metabolic profile should increase the motivation and compliance in the patients, and thereby render better effects.

DETAILED DESCRIPTION:
Patients with overweight or obesity will be recrutied to this open-label, randomized clinical trial. All participants will be informed about the starch- and sucrosereduced diet (SSRD). The diet will be continued for 3 months, with a physical visit with completion of study questionnaires, blood and feces sampling and measurements of anthropometry at baseline, after 6 weeks and 3 months. Thereafter, participants are free to eat whatever they want, but will be examined again after 1 year. Participants will be randomized to whether participants should be informed or not about the metabolic profile measured at week 6. Participants who are randomized to get information about the metabolic profile, will be called when the blood samples have been analysed, and informed about the changes in metabolic and nutrient results between baseline and 6 weeks. The investigators will then evaluate whether participants who were randomized to get information about their blood samples after 6 weeks, will have better compliance to the diet, and thereby have better effect on weight reduction and metabolic profiles. At the blood sampling after 3 months, all participants will be informed about their metabolic profiles. It is also of interest to study the effect at follow-up after 1 year, to see whether participants who were informed at 6 weeks differ from participants who were not.

ELIGIBILITY:
Inclusion Criteria:

* Ålder 18-70 år och språkkunskaper i svenska så att de kan tillgodogöra sig kostinformationen och ifylla formulären.
* BMI ≥25 kg/m2

Exclusion Criteria:

* Allvarlig födoämnesallergi
* Allvarlig hjärt, lung, kardiovaskulär, magtarm, malign eller psykisk sjukdom
* Pågående ätstörning
* Graviditet
* Står redan på en diet såsom vegan diet, regelbunden fasta >15 timmar per dag, eller låg kolhydrat hög fett (LCHF) diet de senaste 3 månaderna
* Alkohol och/eller drogberoende
* Stora ändringar i kroppsvikt de senaste 3 månaderna (≥3 kg)
* Står på viktreducerande läkemedel eller läkemedel som typ GLP-1 analoger

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-12-30 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Mean weight at 3 Months. | 1 year
  All participants are instructed to eat a starch- and sucrosereduced diet (SSRD) during 3 months. Physical meetings are scheduled at baseline, week 6, month 3 and after 1 year, where weight (kg) is measured. Half of the participants are randomized to receive feedback on the metabloic profile after 6 weeks, and the other half will not get any feedback on their blood samples until after 3 months. The hypothesis is that those who recieve feedback on their metabolic profile in the middle of the intervention will be more motivated to follow the diet and be more compliant, which should result in better effects. The reduction in weight from baseline will be calculated. The main outcome is the weight change observed at 3 months.
Change from Baseline in the Mean waist circumference at 3 Months | 1 year
  All participants are instructed to eat a starch- and sucrosereduced diet (SSRD) during 3 months. Physical meetings are scheduled at baseline, week 6, month 3 and after 1 year, where waist circumferense (cm) is measured. Half of the participants are randomized to receive feedback on the metabloic profile after 6 weeks, and the other half will not get any feedback on their blood samples until after 3 months. The hypothesis is that those who recieve feedback on their metabolic profile in the middle of the intervention will be more motivated to follow the diet and be more compliant, which should result in better effects. The reduction in waist circumference from baseline will be calculated. The main outcome is the change observed at 3 months.
Change from Baseline in the body mass composition at 3 Months | 1 year
  All participants are instructed to eat a starch- and sucrosereduced diet (SSRD) during 3 months. Physical meetings are scheduled at baseline, week 6, month 3 and after 1 year, body mass composition is measured. Half of the participants are randomized to receive feedback on the metabloic profile after 6 weeks, and the other half will not get any feedback on their blood samples until after 3 months. The hypothesis is that those who recieve feedback on their metabolic profile in the middle of the intervention will be more motivated to follow the diet and be more compliant, which should result in better effects. The reduction in fat mass from baseline will be calculated. The main outcome is the change observed at 3 months.

SECONDARY OUTCOMES:
The change from baseline in the endocrine profile in blood at 3 months | 1 year
  All participants are instructed to eat a starch- and sucrosereduced diet (SSRD) during 3 months. Physical meetings are scheduled at baseline, week 6, month 3 and after 1 year, where blood samples are collected to measure the endocrine profile. Half of the participants are randomized to receive feedback on the metabolic profile after 6 weeks, and the other half will not get any feedback on their blood samples until after 3 months. The hypothesis is that those who recieve feedback on their metabolic profile in the middle of the intervention will be more motivated to follow the diet and be more compliant, which should result in better effects. The changes in the endocrine profile from baseline will be calculated, where the changes at 3 month will be the main outcome
The change from baseline in the metabolic profile in blood at 3 months | 1 year
  All participants are instructed to eat a starch- and sucrosereduced diet (SSRD) during 3 months. Physical meetings are scheduled at baseline, week 6, month 3 and after 1 year, where blood samples are collected to measure the metabolic profile. Half of the participants are randomized to receive feedback on the metabloic profile after 6 weeks, and the other half will not get any feedback on their blood samples until after 3 months. The hypothesis is that those who recieve feedback on their metabolic profile in the middle of the intervention will be more motivated to follow the diet and be more compliant, which should result in better effects. The changes in metabolic profile from baseline will be calculated, where the changes at 3 month will be the main outcome
The change from baseline in the epigenetic profile measured in blood at 3 months | 1 year
  All participants are instructed to eat a starch- and sucrosereduced diet (SSRD) during 3 months. Physical meetings are scheduled at baseline, week 6, month 3 and after 1 year, where blood samples are collected to measure epigenetics. Half of the participants are randomized to receive feedback on the metabloic profile after 6 weeks, and the other half will not get any feedback on their blood samples until after 3 months. The hypothesis is that those who recieve feedback on their metabolic profile in the middle of the intervention will be more motivated to follow the diet and be more compliant, which should result in better effects. The changes in epigenetic profile from baseline will be calculated, where the changes at 3 month will be the main outcome
The change from baseline in the nutrient profile in blood at 3 months | 1 year
  All participants are instructed to eat a starch- and sucrosereduced diet (SSRD) during 3 months. Physical meetings are scheduled at baseline, week 6, month 3 and after 1 year, where blood samples are collected to measure the nutrient profile. Half of the participants are randomized to receive feedback on the metabloic profile after 6 weeks, and the other half will not get any feedback on their blood samples until after 3 months. The hypothesis is that those who recieve feedback on their metabolic profile in the middle of the intervention will be more motivated to follow the diet and be more compliant, which should result in better effects. The changes in nutrient profile from baseline will be calculated, where the changes at 3 month will be the main outcome
The change from baseline in the inflammatory profile in blood at 3 months | 1 year
  All participants are instructed to eat a starch- and sucrosereduced diet (SSRD) during 3 months. Physical meetings are scheduled at baseline, week 6, month 3 and after 1 year where blood samples are collected to analyse inflammatory parameters. Half of the participants are randomized to receive feedback on the metabloic profile after 6 weeks, and the other half will not get any feedback on their blood samples until after 3 months. The hypothesis is that those who recieve feedback on their metabolic profile in the middle of the intervention will be more motivated to follow the diet and be more compliant, which should result in better effects. The changes in inflammatory profile from baseline will be calculated, where the changes at 3 months will be the main outcome
The change from baseline in the gut microbiota profile measured in feces at 3 months | 1 year
  All participants are instructed to eat a starch- and sucrosereduced diet (SSRD) during 3 months. Physical meetings are scheduled at baseline, week 6, month 3 and after 1 year, where feces samples are collected. Half of the participants are randomized to receive feedback on the metabloic profile after 6 weeks, and the other half will not get any feedback on their blood samples until after 3 months. The hypothesis is that those who recieve feedback on their metabolic profile in the middle of the intervention will be more motivated to follow the diet and be more compliant, which should result in better effects. The changes in gut microbiota profile from baseline will be calculated, where the changes at 3 month will be the main outcome
The change from baseline in the quality of life at 3 months | 1 year
  All participants are instructed to eat a starch- and sucrosereduced diet (SSRD) during 3 months. Physical meetings are scheduled at baseline, week 6, month 3 and after 1 year, where study questionnaires regarding quality of life are completed, and blood and feces samples are collected. Half of the participants are randomized to receive feedback on the metabloic profile after 6 weeks, and the other half will not get any feedback on their blood samples until after 3 months. The hypothesis is that those who recieve feedback on their metabolic profile in the middle of the intervention will be more motivated to follow the diet and be more compliant, which should result in better effects. The changes in quality of life (assessed by HAD, PHQ12-SS, and RAND-36) from baseline will be calculated, where the changes at 3 month will be the main outcome
The change from baseline in bowel symptoms registered by VAS at 3 months | 1 year
  All participants are instructed to eat a starch- and sucrosereduced diet (SSRD) during 3 months. Physical meetings are scheduled at baseline, week 6, month 3 and after 1 year, where study questionnaires regarding bowel symptmos are completed. Bowel symptoms are assessed on visual analog scales (VAS) from 0 mm (no symptoms) to 100 (max symptoms). Half of the participants are randomized to receive feedback on the metabloic profile after 6 weeks, and the other half will not get any feedback on their blood samples until after 3 months. The hypothesis is that those who recieve feedback on their metabolic profile in the middle of the intervention will be more motivated to follow the diet and be more compliant, which should result in better effects. The changes in bowel symptoms from baseline will be calculated, where the changes at 3 month will be the main outcome
The change from baseline in the nutrient intake registered in digital diary food books at 3 months | 1 year
  All participants are instructed to eat a starch- and sucrosereduced diet (SSRD) during 3 months. Physical meetings are scheduled at baseline, week 6, month 3 and after 1 year. Dietary registrations are performed digitally during 3 days at all time points for physical visits. Half of the participants are randomized to receive feedback on the metabloic profile after 6 weeks, and the other half will not get any feedback on their blood samples until after 3 months. The hypothesis is that those who recieve feedback on their metabolic profile in the middle of the intervention will be more motivated to follow the diet and be more compliant, which should result in better effects. The changes in nutrient intake according to the dietary registrations from baseline will be calculated, where the changes at 3 month will be the main outcome
The change from baseline in the inflammatory profile in feces at 3 months | 1 year
  All participants are instructed to eat a starch- and sucrosereduced diet (SSRD) during 3 months. Physical meetings are scheduled at baseline, week 6, month 3 and after 1 year where feces samples are collected to analyse inflammatory parameters. Half of the participants are randomized to receive feedback on the metabloic profile after 6 weeks, and the other half will not get any feedback on their blood samples until after 3 months. The hypothesis is that those who recieve feedback on their metabolic profile in the middle of the intervention will be more motivated to follow the diet and be more compliant, which should result in better effects. The changes in inflammatory profile from baseline will be calculated, where the changes at 3 months will be the main outcome

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Kennbäck, Registered Nurse, Study Chair — Department of Internal Medicine, Skåne University Hospital, 20502 Malmö

IPD SHARING:
Plan to Share IPD: No
Due to ethical rules, it is not allowed to share individual participant data